CLINICAL TRIAL: NCT01928511
Title: SWITCH OR ADD PEGYLATED-INTERFERON IN CHRONIC HEPATITIS B PATIENTS ON LONG TERM NUCLEOS(T)IDE THERAPY (SWAP TRIAL)
Brief Title: Efficacy of Switching or Adding Pegylated Interferon in Chronic Hepatitis B Patients on Long Term Oral Antiviral Therapy
Acronym: SWAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seng Gee Lim (Other)
Collaborators: Tan Tock Seng Hospital (Other); Singapore Clinical Research Institute (Other); Merck Sharp & Dohme LLC (Industry); Singapore General Hospital (Other); Changi General Hospital (Other)
Responsible Party: Sponsor-Investigator, Seng Gee Lim, Director of Hepatology, Dept of Gastroenterology and Hepatology, National University Health System, Singapore
Organization: National University Health System, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MK4031-398; CIRG12may075 (Other Grant/Funding Number: National Medical Research Council Singapore)
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B virus; HBeAg positive; HBeAg negative; antiviral therapy; nucleoside analogues
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — adefovir; entecavir; Tenofovir

STUDY DESIGN:
Intervention Model Description: Three arm parallel study randomised 1:2:2
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continued oral nucleos(t)ide therapy (Active Comparator): Patients assigned to this arm will continue their nucleos(t) analogue
  Interventions: Drug: Nucleos(t)ide analogue therapy
- Add on peg-interferon (Experimental): Patients assigned to this arm will continue their existing nucleos(t)ide therapy and also be assigned peg-interferon alpha 2b 1.5mcg/kg sc weekly
  Interventions: Drug: peg-interferon alpha 2b, 1.5mcg/kg s/c given weekly; Drug: Nucleos(t)ide analogue therapy
- switch to peg-interferon (Experimental): Patients assigned to this arm will stop their existing nucleos(t)ide therapy after one month overlap after starting peg-interferon alpha 2b 1.5mcg/kg sc weekly
  Interventions: Drug: peg-interferon alpha 2b, 1.5mcg/kg s/c given weekly

INTERVENTIONS:
Drug: peg-interferon alpha 2b, 1.5mcg/kg s/c given weekly
  Arms: Add on peg-interferon; switch to peg-interferon
Drug: Nucleos(t)ide analogue therapy
  Other Names: includes lamivudine, adefovir, entecavir, tenofovir or combinations thereof
  Arms: Add on peg-interferon; Continued oral nucleos(t)ide therapy

SUMMARY:
Patients with Chronic Hepatitis B on long term oral antiviral therapy have to continue treatment indefinitely unless they achieve HBeAg seroconversion or HBsAg seroclearance, when therapy can be stopped. While HBeAg seroconversion is a more achievable endpoint, only 20-25% of patients develop this after one year of oral antiviral therapy. HBsAg seroclearance is universally infrequent. Strategies to improve these endpoints such as combination oral antiviral therapy have not been generally successful and recently studies have examined the possibility of switching or adding peginterferon therapy. However these have not been tested adequately in the group of patients that have been on long term oral antiviral therapy. Consequently this study was conceived to evaluate whether switching or adding peginterferon compared to continuing oral antiviral therapy are more efficacious strategies. HBeAg positive and HBeAg negative patients (n=310)will be randomised to continue oral antiviral therapy, switch or add pegylated interferon for 48 weeks in a ratio of 1:2:2 respectively. The study endpoints are HBsAg seroclearance, reduction of qHBsAg >1 log, qHBsAg<200 IU/ml, HBeAg loss and seroconversion, and HBV DNA suppression, all at week 72.

DETAILED DESCRIPTION:
1. HYPOTHESIS AND OBJECTIVES PEG-IFN as an immunomodulatory agent could potentiate the antiviral efficacy of patients on long term nucleos(t)ide analogue therapy and improve early indicators of efficacy, HBeAg loss and reduction in qHBsAg. This study will also test whether add-on compared to switch PEG-IFN is superior, if at all.
2. STUDY DESIGN This is a randomized, open-label, active-controlled study to evaluate safety and the efficacy of HBeAg loss or reduction in qHBsAg >1 log in nucleos(t)ide analogue treated chronic hepatitis B subjects who will be treated with add on PEG (A), switch to PEG (B) or continued nucleos(t)ide analogue (C) for 48 weeks. Patients randomized to Arm B will have a one-month overlap period when switching from existing NA to PEG monotherapy. This is to prevent viral rebound during the switch. Patients will be randomized in a 2:2:1 ratio to one of the 3 treatment arms A, B, and C. Arms A and B are experimental arms. Arm C is the control arm.
3. STUDY POPULATION Approximately 255 subjects will be enrolled into this study.

3.1 Inclusion Criteria

For entry into this study, the following inclusion criteria must be met:

* Age 21 - 70 years old (inclusive)
* Male or female subjects with chronic hepatitis B (ie. presence of positive HBsAg or HBV DNA for at least 6 months.
* On any NA (lamivudine, adefovir, entecavir or tenofovir) for ≥ 1 year
* HBV DNA undetected at screening
* Patient has agreed not to take any other investigational drug or systemic anti-viral, cytotoxic, corticosteroid, immunomodulatory agents or Chinese traditional remedies unless clinically indicated.
* Patient is able to give written consent prior to study start and to comply with the study requirements.
* Women of childbearing age must have a negative urine (ß-HCG) pregnancy test taken within 14 days of starting therapy

3.2 Exclusion Criteria

For entry into this study, the following exclusion criteria must not be met:

* Patient who is on telbivudine.
* Evidence of decompensated liver disease defined as direct (conjugated) bilirubin >1.2xULN, prothrombin time (PT) >1.5x upper limit of normal (ULN), serum albumin <35 g/L, or prior history of clinical hepatic decompensation (egs. ascites, encephalopathy, variceal hemorrhage).
* Evidence of hepatocellular carcinoma.
* Active co-infection with HIV antibody or HCV antibody or HDV antibody positivity.
* Presence of viral resistance defined as virological breakthrough (>1 log increase in HBV DNA from nadir) and presence of viral resistance mutations at the time of screening
* Absolute neutrophil count <1.5 X 109/L or platelets <90 x 109/L or hemoglobin <13 g/dL for men or <12g/dL for women
* Creatinine >1.5 times upper limit of normal or creatinine clearance <60mL/min (performed by central lab)
* Uncontrolled thyroid disease defined as thyroid-stimulating hormone (TSH) >1.2xULN or 0.8xLLN or thyroid dysfunction.
* Any interferon, Immunomodulators, systemic cytotoxic agents, or systemic corticosteroids within 6 months before trial entry.
* Active substance abuse as defined by DSM-IV, Diagnostic Criteria for Drug and Alcohol abuse (appendix 1), which in the opinion of the investigator would make the candidate inappropriate for participation in this study.
* History of clinically relevant psychiatric disease, seizures, central nervous system dysfunction, severe pre-existing cardiac, renal, hematological disease or medical illness that in the investigator's opinion might interfere with therapy.
* History of autoimmune diseases.
* Ophthalmological disorders such as retinopathy, cotton wool spots, optic nerve disorder, retinal hemorrhage, or any other clinically significant abnormality.
* Chronic pulmonary diseases (e.g., chronic obstructive pulmonary disease, interstitial lung disease, pulmonary fibrosis, sarcoidsis).
* Malignant disease within 5 years of trial entry.
* Women who are pregnant and who are not practicing adequate birth control measures, or who are lactating

4.1 Study Treatment

Product, Dose, and Mode of Administration:

Peginterferon α-2b (PEG), 1.5 μg/kg, will be administered weekly by subcutaneous injection for the specified period of time (see Study Design, Arms A and B). Pegintron® (MSD Pharmaceuticals). The dosage will be determined based on the recommended dosing regimen stated in the Pegintron product brochure provided by MSD Pharmaceuticals.

Reference Therapy, Dose, and Mode of Administration:

Patients will be on their existing nucleosid(t)e analogue therapy comprising lamivudine 100mg daily, adefovir 10mg daily, entecavir 0.5mg or 1.0mg daily or tenofovir 300mg daily, (or combinations thereof) all taken as oral medication. These will not be provided by the study protocol.

4.2 Method of Assigning Subjects to a Treatment Randomisation will be performed by computer generated random codes (performed by Singapore Clinical Research Institute) with a masked allocation sequence. Randomization across treatment arms will be stratified by HBeAg status, type of nucleosid(t) analogue, and fibroscan score (<8.8 or ≥8.8) to ensure equal distribution across the 3 treatment groups.

4.3 Blinding/Unblinding There will be no blinding of therapy and the study will be conducted as an open label study as is standard for interferon clinical trials.

5. STUDY ASSESSMENTS AND PROCEDURES 5.1 Time and Event schedule 5.1.1. Screening Visit (Days - 45 to 1) 5.1.2. Baseline Assessments (day 1) 5.1.3. Treatment Assessments (day 2 to week 48) 5.1.4. Pegylated-interferon-free Follow-up (FU) Visits: FU-Week 1 to 24

5.2 Clinical Laboratory Tests Hematology: Full blood count (FBC), prothrombin time and international normalized ratio (PT INR) Chemistry: creatinine, albumin, alkaline phosphatase, aspartate transaminase, alanine transaminase, lactate dehydrogenase, total bilirubin, creatine phosphokinase, alphafetoprotein, (thyroid stimulating hormone and free T4 for patient on PEG-IFN) Urinalysis: Protein, Blood, Glucose Viral serology: HBeAg, anti-HBe, HBsAg, qHBsAg and anti-HBs

6.0 Efficacy assessments HBeAg qualitative Anti-HBe qualitative HBsAg qualitative HBsAg quantitative HBV DNA (real time PCR)

ELIGIBILITY:
Inclusion Criteria:

* Between 21 and 70 years old.
* Documented to be HBsAg positive for ≥ 6 months.
* On any nucleos(t)ide analogue (lamivudine, adefovir, entecavir or tenofovir)for ≥ 1 year
* HBV DNA undetectable by RT PCR at screening
* Patient has agreed not to take any other investigational drug or systemic anti-viral, cytotoxic, corticosteroid, immunomodulatory agents or Chinese traditional remedies unless clinically indicated.
* Patient is able to give written consent prior to study start and to comply with the study requirements.
* Women of childbearing age must have a negative serum (ß-HCG) pregnancy test taken with 14 days of starting therapy

Exclusion Criteria:

* Evidence of decompensated liver disease or hepatocellular carcinoma.
* Have any of the following laboratory tests within 4 weeks of study entry:
* HIV antibody or HCV antibody or HDV antibody positivity
* Absolute neutrophil count < 1.5 X 109/l or platelets < 90 x 109/l or hemoglobin < 13 g/dL for men or 12g/dL for women
* serum albumin <35 g/l or serum bilirubin > 30 mg/l
* creatinine > 1.5 times upper limit of normal
* prothrombin time > 1.5 times control, uncorrected by Vitamin K therapy.
* Any interferon, Immunomodulators, systemic cytotoxic agents, or systemic corticosteroids within 6 months before trial entry.
* Prolonged exposure to known hepatotoxins such as alcohol or drugs.
* History of clinically relevant psychiatric disease, seizures, central nervous system dysfunction, severe pre-existing cardiac, renal, hematological disease or medical illness that in the investigator's opinion might interfere with therapy.
* Malignant disease within 5 years of trial entry.
* Women who are pregnant and who are not practicing adequate birth control measures, or who are lactating

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Reduction in quantitative HBsAg>1 log | Week 72
HBeAg loss | week 72

SECONDARY OUTCOMES:
HBsAg seroclearance | week 72
HBeAg seroconversion | week 72
  In HBeAg positive patients at baseline
HBsAg <200 IU/ml | week 72
undetectable HBV DNA | week 72

CONTACTS AND LOCATIONS:
Overall Officials: Seng Gee Lim, MBBS, FRACP, FRCP, MD, Principal Investigator — National University Health System
Locations (4):
- Singapore (4):
  - Changi General Hospital, Singapore
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

REFERENCES:
- [Derived] Huang DQ, Shen L, Phyo WW, Cloherty G, Butler EK, Kuhns MC, McNamara AL, Holzmayer V, Gersch J, Anderson M, Yang WL, Ngu JH, Chang J, Tan J, Ahmed T, Dan YY, Lee YM, Lee GH, Tan PS, Muthiah M, Khine HTW, Lee C, Tay A, Lim SG. Quantitative HBeAg is a strong predictor of HBeAg loss among patients receiving pegylated interferon. Antiviral Res. 2024 Jul;227:105876. doi: 10.1016/j.antiviral.2024.105876. Epub 2024 Apr 17. PMID 38641023
- [Derived] Lim SG, Yang WL, Ngu JH, Chang J, Tan J, Ahmed T, Dan YY, Lim K, Lee YM, Lee GH, Tan PS, Wai KL, Phyo WW, Khine HHTW, Lee C, Tay A, Chan E. Switching to or Add-on Peginterferon in Patients on Nucleos(t)ide Analogues for Chronic Hepatitis B: The SWAP RCT. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e228-e250. doi: 10.1016/j.cgh.2021.04.031. Epub 2021 Apr 22. PMID 33895361